CLINICAL TRIAL: NCT01038687
Title: Effects of A3309, an Ileal Bile Acid Transport Inhibitor, on Gastrointestinal and Colonic Motor Functions in Female Patients With Functional Constipation
Brief Title: Effect of Ileal Bile Acid Transporter Inhibitor in Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Camilleri, MD (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-006618; UL1RR024150 (NIH)
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Functional Constipation
Keywords: functional constipation; bile acid
MeSH Terms: interventions — elobixibat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A3309 15 mg (Experimental): Patients randomized to this arm received one oral tablet daily of 15 mg A3309 for a period of 14 consecutive days.
  Interventions: Drug: A3309
- A3309 20 mg (Experimental): Patients randomized to this arm received one oral tablet daily of 20 mg A3309 for a period of 14 consecutive days.
  Interventions: Drug: A3309
- Placebo (Placebo Comparator): Patients randomized to this arm received one oral tablet daily of a matching placebo for a period of 14 consecutive days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: A3309 — A3390, a bile acid transport inhibitor was provided in either 15 mg or 20 mg oral tablets
  Other Names: Elobixibat
  Arms: A3309 15 mg; A3309 20 mg
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, parallel group, double-blind, placebo-controlled, dose response, pharmacodynamic and pharmacokinetic study evaluating the effects of A3309 on gastric, intestinal and colonic transit in patients with functional constipation.

DETAILED DESCRIPTION:
Study period Estimated date of first patient enrolled: January 2010 Study design This is a single-center, randomized, parallel group, double-blind, placebo-controlled, dose response, pharmacodynamic and pharmacokinetic study evaluating the effects of A3309 on gastric, intestinal and colonic transit in patients with functional constipation. Doses of 10 or 20 mg A3309 or matching placebo will be administered orally once daily for fourteen (14) consecutive days.

Aim To assess the dose related effects of A3309 on small bowel and overall colonic transit and bowel function in patients with functional constipation.

Number of patients planned Twelve completed female patients with functional constipation in each treatment group for a total of 36 patients.

Diagnosis and main eligibility criteria Female patients with diagnosed functional constipation will be recruited from the local community by public advertisement placed within areas of Mayo Clinic or by a targeted mailing of an informational letter.

Methodology Patients with functional constipation will be screened for eligibility and informed about the study during pre-screening dialogue and also at the initial Visit 1 screen.

Within seven (7) to fourteen (14) days of Visit 1, eligible patients will return for an abbreviated scintigraphy test with images obtained only at 4 and 24 hours following In111 capsule ingestion. A geometric center at 24 hours must be less than or equal to 2.30 to qualify for randomization to study medication. The assigned medication is either 10 or 20 mg A3309 or placebo administered orally once daily for fourteen (14) consecutive days. The allocation to treatment group will be concealed.

A urine pregnancy test will be performed for all females of child bearing potential at Visit 1 and again within the 48 hours prior to the receipt of the isotopes by mouth for both the abbreviated and post-study medication transit scintigraphy tests at Visit 2 and Visit 4. Note that females who are status post-bilateral tubal ligation, hysterectomy or postmenopausal are exempted from this test.

Patients will take study medication at home for eleven (11) consecutive days. Study medication will be administered at the Charlton 7 Clinical Research Unit (CRU) at Visit 4, 5, and 6, the days of scintigraphic assessment of gastric, small bowel and colonic transit of solids performed over a 48 hour period for a total dosing period of fourteen (14) consecutive days.

Within seven (7) to ten (10) days of Visit 6, patients will return to the Charlton 7 CRU for final safety monitoring and an exit physical examination and interview with study staff.

Investigational product, dosage and mode of administration

Patients will take 15 or 20 mg of A3309 or placebo administered orally for eleven (11) consecutive days and report for post-study medication transit scintigraphy on day twelve (12) of dosing. Study medication will be administered once with the In111 capsule on Visit 4 and once immediately before the camera images obtained on Visits 5 and 6. Study medication will be administered at Charlton 7 CRU by a nurse on days 12-14.

Duration of treatment

A3309 or matching placebo will be administered orally once daily for fourteen (14) consecutive days.

Duration of patients' involvement in the study

Each patient will attend seven (7) visits at the clinic during a period of about thirty-one (31) to forty-one (41) days.

Efficacy assessments

* Scintigraphic small bowel and colonic transit
* Assessment of stool frequency and consistency using the Bowel Pattern Diary

Pharmacokinetic analysis Blood samples for analysis of pharmacokinetic (PK) parameters will be collected at Visit 4, before dosing and at 30, 60, 90, 120, 150, 180, 210, and 240 minutes post-dose. PK parameters will be analyzed.

Safety assessments

The following safety assessments will be performed:

* Laboratory safety tests, including a complete blood count (CBC), a comprehensive metabolic panel (CMP), coagulation studies (PT and APTT) and a urinalysis (UA) performed at Visit 1 study entry, Visit 6 completion of transit scintigraphy and final dose of study medication, and Visit 7 study completion. A urine screen for drugs of abuse will be performed once at Visit 1 study entry.
* A 12-lead ECG performed at Visit 1 study entry, Visit 6 completion of post-study medication transit scintigraphy and Visit 7 study completion.
* A physical examination by a study physician at Visit 1 study entry and Visit 7 study completion.
* Vital signs (including temperature, pulse, blood pressure and respiration rate) at every visit
* Urine pregnancy tests performed at Visit 1 study entry and within 48 hours prior to receipt of radiation during the abbreviated transit scintigraphy and post-study medication transit scintigraphy at Visit 2 and Visit 4, respectively
* Interview for concomitant medications and adverse events at every visit

Statistical methods An analysis of covariance (ANCOVA) will be used to compare transit parameters among the treatment groups. The co-variates considered for inclusion in the analyses are age and body mass index (BMI). If necessary a suitable transformation for potential skewness in the distributions of measured volumes may be used (e.g., ANCOVA on ranks or log volumes).

If ANCOVA shows a p value less than or equal to 0.10, then both the 10 mg and 20 mg doses will be compared to placebo (p value less than or equal to 0.025 to correct for 2 pairwise comparisons by Dunnett's Test). Since each of the secondary endpoints assesses a separate hypothesis regarding the effects of A3309, no adjustment in the alpha level for testing multiple types of endpoints is anticipated, and a two-sided significance level of 0.05 will be used in each ANCOVA model.

Statistical Power Based on data acquired using the same methods in the laboratory, the sample size of 12 patients per group provides 80% power to detect differences of approximately 27% to 37% in colonic transit at 24 hours, the primary endpoint. This magnitude of change is considered clinically significant.

PK analyses Plasma concentration vs time curves will be plotted for each subject, on both linear/linear and log10/linear scales. Mean plasma concentration vs time curves will also be presented by dose level. Summary statistics (n, mean, SD, minimum, median, maximum, geometric mean, and coefficient of variation) will be calculated for plasma concentrations at each time point by dose level.

Summary statistics (n, mean, SD, minimum, median, maximum, geometric mean and coefficient of variation) will be presented for all pharmacokinetic parameters by dose level. Geometric mean and coefficient of variation will not be calculated for Tmax. The coefficient of variation will be calculated using the following formula: CV(%) =[exp(SD2)-1]1/2 * 100 where SD=standard deviation of the natural-logarithmically-transformed data.

Analysis data sets The primary analyses will follow the intent to treat (ITT) paradigm with all patients randomized included in the analyses. Those patients with missing response values will have their missing values imputed via the overall (patients with non-missing data) mean and a corresponding adjustment in the ANCOVA residual error variance degrees of freedom (subtracting one for each missing value imputed).

Safety data will be presented for all patients receiving investigational product.

ELIGIBILITY:
INCLUSION CRITERIA

1. Females aged 18 to 65 years old inclusive
2. A diagnosis of functional constipation as defined by two or more of the following:

   1. fewer than three spontaneous complete bowel movements per week
   2. hard or lumpy stools more than 25 % of the time
   3. straining during a bowel movement more than 25 % of the time
3. A normal rectal exam result on file within the past 2 years or performed at screen to exclude the possibility of an evacuation disorder. Examination must exclude findings suggestive of an evacuation disorder such as high sphincter tone at rest, failure of perineal descent and spasm, tenderness or paradoxical contraction of the puborectalis muscles.
4. Females of child-bearing potential (those who have not experienced a bilateral tubal ligation, hysterectomy or menopause) must use an acceptable method of contraception during the study. Acceptable methods are surgical sterilization, hormonal methods such as oral contraceptives, Norplant and Depo-Provera, double barrier method such as a condom and spermicide, and an IUD.

   Abstinent females may participate if they agree to use the double barrier method should they become sexually active during the study.
5. Able to provide written informed consent prior to any study procedures being performed

EXCLUSION CRITERIA

1. Female patients who are pregnant or breast feeding
2. Structural or metabolic diseases/conditions that affect the gastrointestinal system or functional gastrointestinal disorders other than constipation. The long version BDQ will be used to confirm patients have constipation.
3. Unable to withdraw all medications 48 hours prior to Visit 1; any medication that alters GI transit including but not limited to laxatives, magnesium or aluminum-containing antacids. prokinetics, erythromycin, narcotics, anticholinergics, tricyclic antidepressants and SNRIs; analgesic drugs including opiates, NSAIDs, and COX-2 inhibitors (Note: Tylenol is permitted), GABAergic agents and benzodiazepines.

   Note: All other concomitant medications will be reviewed on a case by case basis by the study physicians.
4. Clinical evidence (including but not limited to a clinically significant abnormal physical exam, ECG or laboratory test result in the past medical record) or current clinically significant abnormal physical exam or laboratory test result that could indicate significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other diseases that interfere with the objectives of the study. If a laboratory test result is abnormal and clinically significant, it may be repeated once at the discretion of the PI. If the laboratory test result remains abnormal and clinically significant, the patient will be discontinued from the study and referred to a primary care physician for further evaluation.
5. Patients who are considered by the PI to be alcoholics not in remission or known substance abusers.
6. Patients who have participated in another clinical study in the past 30 days.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Wong BS, Camilleri M, McKinzie S, Burton D, Graffner H, Zinsmeister AR. Effects of A3309, an ileal bile acid transporter inhibitor, on colonic transit and symptoms in females with functional constipation. Am J Gastroenterol. 2011 Dec;106(12):2154-64. doi: 10.1038/ajg.2011.285. Epub 2011 Aug 30. PMID 21876564
- [Derived] Rudling M, Camilleri M, Graffner H, Holst JJ, Rikner L. Specific inhibition of bile acid transport alters plasma lipids and GLP-1. BMC Cardiovasc Disord. 2015 Jul 22;15:75. doi: 10.1186/s12872-015-0070-9. PMID 26197999
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo
Started | 12 | 11 | 13
Completed | 12 | 9 | 12
Not Completed | 0 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 13 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (2.4) | 46.7 (1.9) | 47.5 (2.6) | 44.3 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 13 | 36
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 13 | 36

OUTCOME MEASURES:

1. Primary Outcome: Colonic Transit at 24 Hours
Description: Subjects ingested a Technetium-99m sulfur colloid radiolabeled meal and Indium-111 absorbed on to activated charcoal particles and delivered to the colon by an oral methacrylate-coated capsule. Colonic transit was measured by quantification of radioactive counts via abdominal scintiscans. Overall colonic transit was computed as the colonic geometric center (GC), which is the weighted average of counts in the different colonic regions (ascending, transverse, descending, rectosigmoid and stool), respectively numbered 1 to 5. At any time point, the GC equals the proportion of counts in each colonic region multiplied by its weighting factor: (%ACx1+%TCx2+%DCx3+%RSx4+%stoolx5)/100. As such, a higher GC reflects faster colonic transit. A GC of 1 implies all the isotope is in the ascending colon and a GC of 5 implies all the isotope is in the stool.
Time Frame: 24 hours post-radiolabeled meal
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 13
units on a scale | 2.68 (0.07) | 3.12 (0.07) | 1.93 (0.09)
Statistical Analysis 1: Comparison: A3309 15 mg vs A3309 20 mg vs Placebo; Test type: Superiority; p = 0.059, ANCOVA
Statistical Analysis 2: Comparison: A3309 15 mg vs Placebo; 15mg dose vs placebo; Test type: Superiority; p = 0.18, Dunnett's test
Statistical Analysis 3: Comparison: A3309 20 mg vs Placebo; 20mg dose vs placebo; Test type: Superiority; p = 0.04, Dunnett's test

2. Secondary Outcome: Colonic Filling
Description: Subjects ingested a Technetium-99m sulfur colloid radiolabeled meal and Indium-111 absorbed on to activated charcoal particles and delivered to the colon by an oral methacrylate-coated capsule. Colonic filling was measured by scintigraphy as the percentage of the radiolabeled meal that reached the colon at 6 hours.
Time Frame: 6 hours post-radiolabeled meal
Measure: Mean (Standard Error); unit: percentage of colonic filling
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 13
percentage of colonic filling | 55.8 (9.3) | 60.0 (6.1) | 50.4 (9.6)
Statistical Analysis 1: Comparison: A3309 15 mg vs A3309 20 mg vs Placebo; Test type: Superiority; p = 0.81, ANCOVA
Statistical Analysis 2: Comparison: A3309 15 mg vs Placebo; 15mg dose vs placebo; Test type: Superiority; p = 0.89, Dunnett's test
Statistical Analysis 3: Comparison: A3309 20 mg vs Placebo; 20mg dose vs placebo; Test type: Superiority; p = 0.76, Dunnett's test

3. Secondary Outcome: Gastric Emptying , T1/2
Description: Subjects ingested a Technetium-99m sulfur colloid radiolabeled meal and Indium-111 absorbed on to activated charcoal particles and delivered to the colon by an oral methacrylate-coated capsule. Gastric emptying (GE t 1/2) was measured by scintigraphy and defined as the time required for 50% of the radiolabeled tracer to empty from the stomach.
Time Frame: post-treatment, approximately 12-14 days
Measure: Mean (Standard Error); unit: minutes
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 13
minutes | 165.4 (14.4) | 159.4 (12.8) | 130.8 (5.9)
Statistical Analysis 1: Comparison: A3309 15 mg vs A3309 20 mg vs Placebo; Test type: Superiority; p = 0.075, ANCOVA
Statistical Analysis 2: Comparison: A3309 15 mg vs Placebo; 15mg dose vs placebo; Test type: Superiority; p = 0.058, Dunnett's test
Statistical Analysis 3: Comparison: A3309 20 mg vs Placebo; 20mg dose vs placebo; Test type: Superiority; p = 0.164, Dunnett's test

4. Secondary Outcome: Ascending Colon Emptying t 1/2
Description: Subjects ingested a Technetium-99m sulfur colloid radiolabeled meal and Indium-111 absorbed on to activated charcoal particles and delivered to the colon by an oral methacrylate-coated capsule. Ascending colon emptying t 1/2 was measured by scintigraphy and defined as the time required for 50% of the radiolabeled tracer to empty from the ascending colon.
Time Frame: post-treatment, approximately 12-14 days
Measure: Mean (Standard Error); unit: hours
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 13
hours | 14.0 (3.6) | 5.8 (1.9) | 14.8 (1.6)
Statistical Analysis 1: Comparison: A3309 15 mg vs A3309 20 mg vs Placebo; Test type: Superiority; p = 0.084, ANCOVA
Statistical Analysis 2: Comparison: A3309 15 mg vs Placebo; 15mg vs placebo; Test type: Superiority; p = 0.98, Dunnett's test
Statistical Analysis 3: Comparison: A3309 20 mg vs Placebo; 20mg vs placebo; Test type: Superiority; p = 0.079, Dunnett's test

5. Secondary Outcome: Colonic Transit at 8 Hours
Description: as for outcome 1
Time Frame: 8 hours post-radiolabeled meal
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 13
units on a scale | 1.98 (0.55) | 2.82 (0.55) | 1.20 (0.09)
Statistical Analysis 1: Comparison: A3309 15 mg vs A3309 20 mg vs Placebo; Test type: Superiority; p = 0.058, ANCOVA
Statistical Analysis 2: Comparison: A3309 15 mg vs Placebo; 15mg dose vs placebo; Test type: Superiority; p = 0.32, Dunnett's test
Statistical Analysis 3: Comparison: A3309 20 mg vs Placebo; 20mg dose vs placebo; Test type: Superiority; p = 0.034, Dunnett's test

6. Secondary Outcome: Colonic Transit at 48 Hours
Description: as for outcome 1
Time Frame: 48 hours post-radiolabeled meal
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 13
units on a scale | 3.64 (0.07) | 3.91 (0.07) | 2.18 (0.09)
Statistical Analysis 1: Comparison: A3309 15 mg vs A3309 20 mg vs Placebo; Test type: Superiority; p = 0.001, ANCOVA
Statistical Analysis 2: Comparison: A3309 15 mg vs Placebo; 15mg dose vs placebo; Test type: Superiority; p = 0.002, Dunnett's test
Statistical Analysis 3: Comparison: A3309 20 mg vs Placebo; 20mg vs placebo; Test type: Superiority; p = 0.001, Dunnett's test

7. Secondary Outcome: Stool Frequency
Description: Subjects maintained a validated daily bowel diary and recorded the number of bowel movements each day during treatment.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: bowel movements
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 13
bowel movements | 1.33 (0.15) | 2.14 (0.39) | 1.43 (0.24)
Statistical Analysis 1: Comparison: A3309 15 mg vs A3309 20 mg vs Placebo; Test type: Superiority; p = 0.091, ANCOVA
Statistical Analysis 2: Comparison: A3309 15 mg vs Placebo; 15mg dose vs placebo; Test type: Superiority; p = 0.99, Dunnett's test
Statistical Analysis 3: Comparison: A3309 20 mg vs Placebo; 20mg vs placebo; Test type: Superiority; p = 0.103, Dunnett's test

8. Secondary Outcome: Stool Consistency
Description: Subjects maintained a validated daily bowel diary during treatment and recorded stool consistency according to the Bristol Stool Form Scale, where: 1= separate hard lumps; 2= lumpy sausage-shape; 3= cracked sausage; 4= smooth and soft sausage; 5=soft blobs; 6=mushy, fluffy pieces; 7= watery, no solid pieces.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 13
units on a scale | 4.17 (0.32) | 4.42 (0.32) | 2.69 (0.24)
Statistical Analysis 1: Comparison: A3309 15 mg vs A3309 20 mg vs Placebo; Test type: Superiority; p = 0.001, ANCOVA
Statistical Analysis 2: Comparison: A3309 15 mg vs Placebo; 15mg dose vs placebo; Test type: Superiority; p = 0.002, Dunnett's test
Statistical Analysis 3: Comparison: A3309 20 mg vs Placebo; 20mg dose vs placebo; Test type: Superiority; p = 0.001, Dunnett's test

9. Secondary Outcome: Treatment Effectiveness of A3309
Description: Subject perception of treatment efficacy was measured using a 5 point numerical scale where 1=not at all effective to 5=extremely effective.
Time Frame: Day 14
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 13
score on a scale | 3.7 (0.3) | 2.4 (0.4) | 4.3 (0.3)
Statistical Analysis 1: Comparison: A3309 15 mg vs A3309 20 mg vs Placebo; Test type: Superiority; p = 0.002, ANCOVA
Statistical Analysis 2: Comparison: A3309 15 mg vs Placebo; 15mg dose vs placebo; Test type: Superiority; p = 0.053, Dunnett's test
Statistical Analysis 3: Comparison: A3309 20 mg vs Placebo; 20mg dose vs placebo; Test type: Superiority; p = 0.002, Dunnett's test

ADVERSE EVENTS:
Time Frame: Adverse events were collected on each subject from enrollment until 7-10 days after the last day of the study medication, for approximately one month.
Arm/Group | A3309 15 mg | A3309 20 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 12/12 | 11/11 | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A3309 15 mg (N=12) | A3309 20 mg (N=11) | Placebo (N=13)
Abdominal cramps/pain (Gastrointestinal disorders) | 4 (4) | 6 (6) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Borboygmi (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Stomach upset (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hemorrhoid pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation exacerbation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bloating (General disorders) | 0 (0) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stress (General disorders) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (General disorders) | 0 (0) | 0 (0) | 4 (4)
Headache (General disorders) | 0 (0) | 0 (0) | 10 (10)
Lightheadness (General disorders) | 0 (0) | 0 (0) | 2 (2)
Lethargy (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Body ache (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2010-06-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT01038687/Prot_SAP_ICF_000.pdf